CLINICAL TRIAL: NCT06792292
Title: Real-World Experience of Artificial Intelligence-Assisted Colonoscopy in Colorectal Cancer Screening in a General Hospital: A Single-Center Cohort Phase IV Study
Brief Title: Artificial Intelligence-Assisted Colonoscopy in Colorectal Cancer Screening in a General Hospital
Acronym: Delta-AI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chirec (Other)
Responsible Party: Principal Investigator, Erik Francois, Principal Investigator, Chirec
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024 Chirec Delta Colo-AI
Record Dates: First submitted 2025-01-12; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Artificial Intelligence; Colonic Adenoma; Colonic Neoplasms; Colonic Polyp; Colonoscopy
Keywords: colo-rectal cancer screening; artificial intelligence assisted colonoscopy
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps

STUDY DESIGN:
Intervention Model Description: Arm 1- Conventional colonoscopy Arm 2- Colonoscopy assisted by artificial intelligence system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CCP: conventional colonoscopy procedure (Active Comparator): The conventional colonoscopy arm subjects will undergo a screening colonoscopy without assistance from artificial intelligence.
  Interventions: Other: conventional colonoscopy procedure
- ACP: artificial intelligence-assisted colonoscopy procedure (Active Comparator): The artificial intelligence-assisted colonoscopy arm subjects will undergo a screening colonoscopy with assistance from an artificial intelligence module.
  Interventions: Other: artificial intelligence-assisted colonoscopy procedure

INTERVENTIONS:
Other: conventional colonoscopy procedure — Study subjects in this interventional arm will undergo conventional colonoscopy.
  Arms: CCP: conventional colonoscopy procedure
Other: artificial intelligence-assisted colonoscopy procedure — Study subjects in this interventional arm will undergo colonoscopy done with a commercially-available module that uses artificial intelligence to highlight suspected polyps on the screen during colonoscopy. This module also attempts to characterize the detected polyp as adenomatous or not. The detection and characterization of polyps is in real time, during the procedure.
  Arms: ACP: artificial intelligence-assisted colonoscopy procedure

SUMMARY:
Cancer can develop in the colon, or large bowel. Examination of the colon with a tube fitted with a camera is called a colonoscopy.

Colonoscopy allows detection of small growths in the colon, called "polyps". Polyps can often be removed during colonoscopy. Some of these polyps are called adenomas and can become cancer after several years.

A good colonoscopy aims to find and take out as many of these polyps as possible.

A quality indication of colonoscopy is the "adenoma detection rate" (ADR). It should be high, meaning many polyps are detected and taken out.

New artificial intelligence devices to assist colonoscopy seem to increase the ADR, and maybe help prevent cancer even better than normal colonoscopy.

The goal of this clinical trial is to compare the ADR when using standard colonoscopy to the ADR with artificial intelligence (AI)-assisted colonoscopy.

DETAILED DESCRIPTION:
The colon is a part of the bowel where colon cancer can develop.

It is possible to prevent colon cancer by doing a screening test called a colonoscopy.

The colonoscopy procedure allows detection of "polyps" which can often be removed during the procedure. Some of these polyps are called adenomas and can become cancer after several years.

A good colonoscopy aims to find and take out as many of these polyps as possible.

A quality indication of colonoscopy is the "adenoma detection rate" (ADR). It should be high, meaning many polyps are detected and taken out.

New artificial intelligence devices to assist colonoscopy seem to increase the ADR, and maybe help prevent cancer even better than normal colonoscopy.

The goal of this clinical trial is to compare the ADR when using standard colonoscopy to the ADR with artificial intelligence (AI)-assisted colonoscopy.

Patients who are scheduled to have screening colonoscopy and who agree to participate, and are aged 45 years or more, will be randomly assigned to receive either standard colonoscopy or AI-assisted colonoscopy.

The main objective of this study is the difference in the ADR between a conventional colonoscopy procedure and an AI-assisted colonoscopy procedure.

Secondary objectives will compare the 2 groups (conventional colonoscopy and AI-assisted colonoscopy) regarding polyp size, polyp quantity, polyp histology (laboratory analysis of the polyp that was taken out), polyp dysplasia grade (how close the polyp is to cancer), polyp location in the colon, endoscopist experience (older or younger doctor), time of day and colonoscopy preparation quality (how clean the bowel is).

With these results we can show that AI-assisted colonoscopy is useful or not to help better prevent colon cancer.

ELIGIBILITY:
Inclusion criteria:

* Patient (woman or man) candidate for a screening colonoscopy - Age: 45 to 74 years included
* Absence of inflammatory bowel disease
* Absence of significant digestive symptoms indicating colonoscopy (i.e. screening is the only indication for the examination)
* Patient able to understand the concept of the study and agreeing to participate

Exclusion criteria:

* Patient outside the inclusion age
* All exclusion criteria for a colonoscopy.
* The indication for colonoscopy is not simple screening; for example, assessment of anemia, rectal bleeding, weight loss or abdominal pain.
* Patient's refusal to participate, or patient's inability to understand the study concept
* Any patient with major psychological or psychiatric disorders.

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 765 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Adenoma Detection Rate in Conventional versus Artificial Intelligence-Assisted Colonoscopy | 1 day
  The main objective of this study is the difference in the detection rate of colorectal adenomas in individuals over 45 years old during colonoscopies for colon cancer screening between a conventional colonoscopy procedure (CCP) and a colonoscopy procedure with AI (ACP).

SECONDARY OUTCOMES:
The difference in the detection rate of colorectal adenomas according to size by group (5 mm/6-9 mm/>10 mm) between a conventional colonoscopic procedure (CCP) and a colonoscopy procedure with AI (ACP). | 1 day
  Detection rate of diminutive, small, and large polyps will be compared between a conventional colonoscopic procedure (CCP) and a colonoscopy procedure with AI (ACP).
The difference in the detection rate of colorectal adenomas according to the number per group (n=1-2/n= 3-10/n >10) between a conventional colonoscopic procedure (CCP) and a colonoscopy procedure with AI (ACP). | 1 day
  The number of adenomas detected during the procedure will be compared between a conventional colonoscopic procedure (CCP) and a colonoscopy procedure with AI (ACP).
The difference in the detection rate of colorectal adenomas based on histology by group (hyperplastic/conventional adenomas/serrated adenomas/adenocarcinoma) between a conventional colonoscopic procedure (PCC) and a colonoscopy procedure with AI. | 1 month
  Adenomas have different histologic types. After obtaining histology, the detection rate of the various histologic types will be compared between a conventional colonoscopic procedure (CCP) and a colonoscopy procedure with AI (ACP).
The difference in detection rate of colorectal adenomas based on dysplastic grade by group | 1 day
  The difference in detection rate of colorectal adenomas based on dysplastic grade
  by group (conventional or serrated adenomas/low-grade dysplasia/high-grade dysplasia/adenocarcinoma) or Narrow Band Imaging International Colorectal Endoscopic (NICE) (stages 1, 2 or 3) classification or Japan Narrow Band Imaging Expert Team (JNET) classification (stages 1, 2A and 2B, or 3) between a conventional colonoscopy procedure (CCP) and a colonoscopy procedure with AI (ACP).
The difference in the detection rate of colorectal adenomas depending on the location by group (rectum/left colon/transverse colon/right colon) between a conventional colonoscopic procedure (CCP) and a colonoscopy procedure with AI (ACP). | 1 day
  Location of adenomas will be compared between a conventional colonoscopic procedure (CCP) and a colonoscopy procedure with AI (ACP).
The difference in the detection rate of colorectal adenomas according to experience by group of colonoscopists | 1 day
  The difference in the detection rate of colorectal adenomas according to experience by group (Colonoscopists aged 45-55 years/56-65 years/>66 years) between a conventional colonoscopic procedure (CCP) and a conventional colonoscopic procedure (CCP) colonoscopy with AI (ACP).
The difference in the detection rate of colorectal adenomas depending on the time of day . | 1 day
  The difference in the detection rate of colorectal adenomas depending on the time of day (before 11:00/between 11:00 and 15:00/after 15:00) and the number of colonoscopies (Colonoscopy from 1 to 6 per half-day) per group (hyperplastic/conventional adenomas/scalloped adenomas/adenocarcinoma) between a conventional colonoscopic procedure (PCC) and a colonoscopy procedure with AI (ACP).
The difference in the detection rate of colorectal adenomas according to colonic preparation by group (Boston Score 9/6-8/<6) between a conventional colonoscopic procedure (PCC) and a colonoscopy procedure with AI (ACP). | 1 day
  The difference in the adenoma detection rate according to the quality of colonic preparation will be compared between a conventional colonoscopic procedure (CCP) and a colonoscopy procedure with AI (ACP).

CONTACTS AND LOCATIONS:
Overall Officials: Denis Franchimont, M.D., PhD, Study Chair — Chirec
Locations (1):
- Hopital Delta Chirec, Auderghem, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data will include anonymized demographic information, clinical outcomes, laboratory results, and recorded adverse events.
  Access to the data will be available to qualified researchers, with requests submitted by contacting one of the investigators.
  The investigators will employ strict data protection measures, ensuring all shared data is de-identified and in compliance with applicable data protection laws. Access to the individual participant data will be contingent on the signing of a data sharing agreement that outlines the intended use of the data and adherence to ethical guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The investigators anticipate that data will be available within six months after the completion of the trial and publication of the primary findings, and for a period of one year thereafter.
Access Criteria: Access to the data will be available to qualified researchers, with requests submitted by contacting one of the investigators.

REFERENCES:
- [Background] Spadaccini M, Marco A, Franchellucci G, Sharma P, Hassan C, Repici A. Discovering the first US FDA-approved computer-aided polyp detection system. Future Oncol. 2022 Apr;18(11):1405-1412. doi: 10.2217/fon-2021-1135. Epub 2022 Jan 27. PMID 35081745
- [Background] Repici A, Badalamenti M, Maselli R, Correale L, Radaelli F, Rondonotti E, Ferrara E, Spadaccini M, Alkandari A, Fugazza A, Anderloni A, Galtieri PA, Pellegatta G, Carrara S, Di Leo M, Craviotto V, Lamonaca L, Lorenzetti R, Andrealli A, Antonelli G, Wallace M, Sharma P, Rosch T, Hassan C. Efficacy of Real-Time Computer-Aided Detection of Colorectal Neoplasia in a Randomized Trial. Gastroenterology. 2020 Aug;159(2):512-520.e7. doi: 10.1053/j.gastro.2020.04.062. Epub 2020 May 1. PMID 32371116
- [Background] Gupta S, Lieberman D, Anderson JC, Burke CA, Dominitz JA, Kaltenbach T, Robertson DJ, Shaukat A, Syngal S, Rex DK. Recommendations for Follow-Up After Colonoscopy and Polypectomy: A Consensus Update by the US Multi-Society Task Force on Colorectal Cancer. Gastrointest Endosc. 2020 Mar;91(3):463-485.e5. doi: 10.1016/j.gie.2020.01.014. Epub 2020 Feb 7. No abstract available. PMID 32044106
- [Background] Kaminski MF, Thomas-Gibson S, Bugajski M, Bretthauer M, Rees CJ, Dekker E, Hoff G, Jover R, Suchanek S, Ferlitsch M, Anderson J, Roesch T, Hultcranz R, Racz I, Kuipers EJ, Garborg K, East JE, Rupinski M, Seip B, Bennett C, Senore C, Minozzi S, Bisschops R, Domagk D, Valori R, Spada C, Hassan C, Dinis-Ribeiro M, Rutter MD. Performance measures for lower gastrointestinal endoscopy: a European Society of Gastrointestinal Endoscopy (ESGE) quality improvement initiative. United European Gastroenterol J. 2017 Apr;5(3):309-334. doi: 10.1177/2050640617700014. Epub 2017 Mar 16. PMID 28507745
- [Background] Hassan C, Antonelli G, Dumonceau JM, Regula J, Bretthauer M, Chaussade S, Dekker E, Ferlitsch M, Gimeno-Garcia A, Jover R, Kalager M, Pellise M, Pox C, Ricciardiello L, Rutter M, Helsingen LM, Bleijenberg A, Senore C, van Hooft JE, Dinis-Ribeiro M, Quintero E. Post-polypectomy colonoscopy surveillance: European Society of Gastrointestinal Endoscopy (ESGE) Guideline - Update 2020. Endoscopy. 2020 Aug;52(8):687-700. doi: 10.1055/a-1185-3109. Epub 2020 Jun 22. PMID 32572858
- [Background] Brenner H, Hoffmeister M, Stegmaier C, Brenner G, Altenhofen L, Haug U. Risk of progression of advanced adenomas to colorectal cancer by age and sex: estimates based on 840,149 screening colonoscopies. Gut. 2007 Nov;56(11):1585-9. doi: 10.1136/gut.2007.122739. Epub 2007 Jun 25. PMID 17591622
- [Background] Saftoiu A, Hassan C, Areia M, Bhutani MS, Bisschops R, Bories E, Cazacu IM, Dekker E, Deprez PH, Pereira SP, Senore C, Capocaccia R, Antonelli G, van Hooft J, Messmann H, Siersema PD, Dinis-Ribeiro M, Ponchon T. Role of gastrointestinal endoscopy in the screening of digestive tract cancers in Europe: European Society of Gastrointestinal Endoscopy (ESGE) Position Statement. Endoscopy. 2020 Apr;52(4):293-304. doi: 10.1055/a-1104-5245. Epub 2020 Feb 12. PMID 32052404
- [Background] Hassan C, Spadaccini M, Iannone A, Maselli R, Jovani M, Chandrasekar VT, Antonelli G, Yu H, Areia M, Dinis-Ribeiro M, Bhandari P, Sharma P, Rex DK, Rosch T, Wallace M, Repici A. Performance of artificial intelligence in colonoscopy for adenoma and polyp detection: a systematic review and meta-analysis. Gastrointest Endosc. 2021 Jan;93(1):77-85.e6. doi: 10.1016/j.gie.2020.06.059. Epub 2020 Jun 26. PMID 32598963